CLINICAL TRIAL: NCT06511765
Title: Anesthetic Block of the Erector Muscles of the Lumbar Spine to Relieve Acute Lumbar Pain: Pilot Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLOCLOMB
Record Dates: First submitted 2024-07-03; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Lumbago
Keywords: anesthetic blocks; pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous injection of Ropivacaine combined with Dexamethasone + usual treatment (Experimental): The experimental treatment consists in one single interlaminal injection of 2x20ml Ropivacaine (0.375%) distributed over the L4-L5 (Lumbar vertebrae 4 and 5) and L5-S1 (Lumbar vertebrae 5 and sacrum 1) levels on both sides, combined with 2x4ml Dexamethasone soluble (i.e. 2x1ml). This dose and method of administration are those required for locoregional anesthesia.
  Interventions: Drug: Ropivacaine and dexamethasone injection solution
- Intravenous injection of Placebo (sodium chloride 0.9%) + usual treatment (Placebo Comparator): The placebo treatment consists in one single interlaminal injection of 2x20ml sodium chloride 0.9% distributed over the L4-L5 and L5-S1 levels on both sides.
  Interventions: Drug: Sodium Chloride 0.9% Injection Solution

INTERVENTIONS:
Drug: Ropivacaine and dexamethasone injection solution — Injection of Ropivacaine and dexamethasone
  Arms: Intravenous injection of Ropivacaine combined with Dexamethasone + usual treatment
Drug: Sodium Chloride 0.9% Injection Solution — Injection of sodium chloride 0.9%
  Arms: Intravenous injection of Placebo (sodium chloride 0.9%) + usual treatment

SUMMARY:
This study concerns the treatment of recent lumbago and aims to evaluate the efficacy of an anesthetic block of the erector spinae muscles combining ropivacaine and dexamethasone. This treatment is routinely used in several institutions in France, but has never been the subject of a randomized placebo-controlled study to assess its efficacy at D4 of treatment.

The BLOCLOMB comparative, randomized, double-blind study aims to validate the efficacy, over the first 4 days, of anesthetic blocks of the erector spinae muscles, during recent lumbago, on the pain of muscular contractures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with lumbago lasting less than 7 days despite analgesic / NSAID treatment.
2. Patient with NS pain > 6
3. Patient with Oswestry score > or equal to 30
4. Patient informed of the trial and having signed the informed consent form prior to any trial-specific procedure,
5. Patient willing and able to undergo all planned examinations and procedures in compliance with the clinical trial protocol,
6. Patient affiliated to a social security or any health insurance.

Exclusion Criteria:

1. Presence of "red flag" (non-disc lumbago):

   * Motor deficit or signs of horsetail irritation
   * Inflammatory pain waking up in the 2nd half of the night
   * Tumoral context
   * Infectious context or fever
   * Altered general condition
   * Traumatic context
   * Osteoporotic context
2. Risk of infection
3. Patient with poor local skin condition
4. Patient on AVK or anti-Xa anticoagulation, or bleeding disorder (antiaggregants authorized)
5. Patients with hypersensitivity to Ropivacaine or any of its excipients: Sodium chloride, hydrochloric acid sodium hydroxide
6. Patient with sciatica
7. Patient with chronic respiratory insufficiency
8. Patient with cardiac rhythm disorders
9. Pregnant or breastfeeding woman or woman refusing effective contraception
10. Patient deprived of liberty or under legal protection (guardianship or curator)
11. Patient participating in another clinical research protocol involving a drug or medical device
12. Patient unable to follow the protocol, as judged by the investigator
13. Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Lumbar pain in activity | At Hour 0-Hour1-Hour4-Hour8-Hour12 and Day 1-Day2-Day3-Day4. (Hour 0=injection time, Day 1=One day after injection time)
  Area under the curve of lumbar pain in activity measured by the patient on a numeric scale (from 0=no pain, and 10=unbearable pain)

SECONDARY OUTCOMES:
Consumption of concomitant lumbago treatments | From Day 0 (day of injection) to Day 4
  Recording of analgesics and NSAIDs, physiotherapy, manipulations, open surgery, etc
Lumbar pain at rest | Day 4
  Lumbar pain measured by the patient on a numeric scale
Lumbar pain in activity | Day 4
  Lumbar pain measured by the patient on a numeric scale
Lumbar pain at rest | At Hour 0-Hour1-Hour4-Hour8-Hour12 and Day 1-Day 2-Day 3-Day 4-Day 7-Day 14-Day 21-Day 28
  Area under the curve of lumbar pain at rest measured by the patient on a numeric scale
Lumbar Pain < 3 | Day 4
  Percentage of patients with pain < 3 (measured by the patient on a numeric scale, at rest)
Algofunctional index | Day 0, Day 4 and Day 28
  Oswestry questionnaire: comprises 10 questions on pain, personal care, load-bearing, walking, sitting, standing, sleep, sex life, social life and travel. Each question offers 6 answers, with a score from 0 to 6, which the patient must choose; a score of 0 corresponds to normal function, and a score of 6 to severely impaired function.
  The score obtained is multiplied by 2 to obtain a percentage of disability, with 0% for no disability, and 100% for the greatest disability.
Duration of the interruption of current activities | 28 days
  Number of days without current activities
Duration of the interruption of work | 28 days
  Number of days of sick leave
Complications | 28 days
  Complications will focus on the following adverse events:
  1. injection-site hematoma, nerve damage, limb pain, convulsions, respiratory discomfort, bradycardia, severe vagal malaise
  2. fall, iatrogenic infection
  3. new lumbago, sciatica or complicated crural neuralgia (neurological deficit, cauda equina syndrome)
  4. allergy, digestive complication, renal complication
  5. other to be specified

CONTACTS AND LOCATIONS:
Locations (1):
- Santé Atlantique ELSAN, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No